CLINICAL TRIAL: NCT03540225
Title: Vaginal Progesterone for the Prevention of Preterm Birth in Twins: A Pilot Randomised, Factorial Designed Trial (POPPET)
Brief Title: Vaginal Progesterone for the Prevention of Preterm Birth in Twins
Acronym: POPPET
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Fail to sort out the logistics of study drugs due to funding problems
Sponsor: Chiu Yee Liona Poon (Other)
Responsible Party: Sponsor-Investigator, Chiu Yee Liona Poon, Associate Professor (Clinical), Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2016.594-T
Record Dates: First submitted 2018-05-07; First posted 2018-05-30 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Premature Birth; Twin Pregnancy
Keywords: Progesterone
MeSH Terms: conditions — Premature Birth | interventions — Progesterone; Utrogestan

STUDY DESIGN:
Intervention Model Description: 2 x 2 factorial designed trial with two factors of 200mg vs. 400mg vaginal progesterone daily from 11-14 weeks' gestation vs. 20-24 weeks'
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Early Low-dose Arm (Experimental): Start from 11-14 week: 200 mg self-administered vaginal progesterone daily
  Interventions: Drug: Progesterone
- Early High-dose Arm (Experimental): Start from 11-14 week: 400 mg self-administered vaginal progesterone daily
  Interventions: Drug: Progesterone
- Late Low-dose Arm (Experimental): Start from 20-24 week: 200 mg self-administered vaginal progesterone daily
  Interventions: Drug: Progesterone
- Late High-dose Arm (Experimental): Start from 20-24 week: 400 mg self-administered vaginal progesterone daily
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — Utrogestan Vaginal 200 mg or 400 mg daily from 11-14 Week or 20-24 Week until 34 Week
  Other Names: Utrogestan

SUMMARY:
This trial is a randomised, multi-centre, 2 x 2 factorial designed pilot trial with two factors of 200mg vs. 400mg progesterone self-administered daily from 11-14 weeks' gestation vs. 20-24 weeks' gestation, to compare the median gestational age (in days) at delivery between the comparison groups.

DETAILED DESCRIPTION:
Randomised studies in singleton pregnancies suggest that the risk of preterm birth can be decreased by using of progesterone. However, in twin pregnancies, no significant reduction in preterm birth has been demonstrated in any trial.

One explanation for the lack of benefit of progesterone in previous twin studies may result from a suboptimal dosage. The investigators therefore hypothesize that progesterone dosages that are sufficient for singleton pregnancies are insufficient for twins and this is likely to be one of the reasons why prophylactic progesterone has failed to reduce preterm birth in twins.

Another possible explanation for the negative findings in previous twin studies may result from administration beginning too late in the second-trimester. It is thought that the mechanism of preterm birth in twin pregnancies is more strongly related to exaggerated uterine distension, which may override any benefit of progesterone on the cervix after a threshold has been reached. It is also plausible that cervical shortening occurs earlier in twin pregnancies than with singletons, and that treatment is required before a threshold of shortening is reached or before any inflammation-mediated component to the initiation of preterm birth has been established as the biological mechanisms by which preterm birth occurs differ from those in singleton pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Dichorionic diamniotic (DCDA) pregnancies
* Live fetuses at 11-13 weeks of gestation,
* Informed and written consent

Exclusion Criteria:

* High-risk for aneuploidies,
* Pregnancies complicated by major fetal abnormality identified at the 11-13 weeks or 20-24 weeks assessment,
* Hypersensitivity to progesterone,
* Women taking progesterone regularly or at any time within the previous 7 days,
* Concurrent participation in another drug trial or at any time within the previous 28 days,
* Women who are unconscious or severely ill, those with learning difficulties, or serious mental illness,
* Any other reason the clinical investigators think will prevent the potential participant from complying with the trial protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The median gestational age (in days) at delivery | At delivery

SECONDARY OUTCOMES:
The incidence of spontaneous preterm birth | Less than 34 weeks (237 days) of gestation
Birth weight | At delivery
Stillbirth or neonatal death due to any cause | At delivery
Major adverse outcomes before discharge from the hospital | Within the first year
  Intraventricular hemorrhage, respiratory distress syndrome, retinopathy of prematurity, or necrotizing entercolitis.
Need for neonatal special care | Between birth and 28 days of age
  Admission to a neonatal intensive care unit, ventilation, phototherapy, treatment for proven or suspected sepsis, or blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Liona CY Poon, MD, Principal Investigator — Chinese University of Hong Kong
Locations (4):
- Hong Kong (4):
  - Kwong Wah Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No